CLINICAL TRIAL: NCT02681289
Title: Physiotherapy of At-Risk Infants, Physiotherapist or Family? A Randomized Intervention Study
Brief Title: Physiotherapy of At-Risk Infants, Physiotherapist or Family?
Acronym: Infant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Nilay Comuk Balci, Pt, PhD, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO13 186-01
Record Dates: First submitted 2016-02-07; First posted 2016-02-12 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Problem With Growth of an Infant
Keywords: infant; risk; rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- physiotherapy group (Experimental): Early goal directed neuromotor therapy applied by physiotherapist
  Interventions: Other: Early goal directed neuromotor therapy
- family group (Experimental): Early goal directed neuromotor therapy applied by family
  Interventions: Other: Early goal directed neuromotor therapy

INTERVENTIONS:
Other: Early goal directed neuromotor therapy — Early goal directed neuromotor therapy (NGDT) is referred to as 'task-oriented' and is built on contemporary system theories of motor control. The development and learning of new skills occur in an interaction between the child, the task to be performed and the particular environment in which the activity takes place.

SUMMARY:
Early physiotherapy reduces neuromotor problems in at-risk infants. This study was planned to compare the effects of an early goal-directed neuromotor physiotherapy (GDNT) application between preterm and term at-risk infants.

DETAILED DESCRIPTION:
Early physiotherapy reduces neuromotor problems in at-risk infants. This study was planned to compare the effects of an early goal-directed neuromotor physiotherapy (GDNT) application between preterm and term at-risk infants. Eighteen at-risk infants between the ages of 0 and 12 months were assigned to the preterm and term groups according to their gestational and corrected age. Each group received GDNT for 45 min, three days per week for 12 weeks. The effectiveness of the therapy was measured using Alberta Infant Motor Scale (AIMS), Hammersmith Infant Neurological Examination (HINE), and Goal Attainment Scale (GAS).

ELIGIBILITY:
Inclusion Criteria:

* being diagnosed as "at-risk" by a pediatric neurologist, having intraventricular hemorrhage, periventricular leucomalacia, hypoxic ischemic encephalopathy, and prematurity, Apgar score of 5 or less at 5 min, chronic lung disease, seizures, meningitis, hyperbilirubinemia, being twins or triplets, and having intrauterine growth restriction;
* being outside of the neonatal intensive care unit;
* being between 0 and 12 months old (corrected age for premature infants);
* having a family acceptance for the participation in 12 weeks of therapy program.

Exclusion Criteria:

* having congenital anomalies, musculoskeletal disorders, cyanotic congenital heart disease and mechanical dependency, and
* lack of informed content by the parents.

Max Age: 15 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Hammersmith Infant Neurological Examination (HINE) | 12 weeks
  It includes three sections, the Neurological Examination, the Development of Motor Functions and the State of Behaviour.The data obtained in the second and third sections are not included in the calculation of global optimality scores. The overall score ranges from a minimum of 0 to a maximum of 78. At 9 or 12 months, the scores equal or above 73 are regarded as optimal, if below 73 as sub-optimal; while at 3 and 6 months healthy term infants scored equal or above 67 and 70 (median) respectively.
Alberta Infant Motor Scale (AIMS) | 12 weeks
  This scale is a norm-referenced observational tool designed for the evaluation of gross motor development in infants from birth to 18 months of age or the acquisition of independent walking. It consists of 58 items and four subscales: supine (9 items), prone (21 items), sitting (12 items) and standing (16 items), which are observed in postural alignment, antigravity movements and surface contact.The obtained score (0-60 points) was converted to a normative age-dependent percentile rank (5th,10th,25th, 50th, 75th or 90th percentiles). A score less than the 10th percentile was classified as possibly delayed motor development.
Goal Attainment Scale (GAS) | 12 weeks
  GAS methods required practitioners to set rehabilitation goals in collaboration with the client and family. or significant others, such as a carer. For each goal, the client and practitioner developed detailed and very specific observable and quantifiable descriptions of possible outcomes Five outcome levels were identified,including the expected or desired level of performance or outcome, 2 levels that would be seen as less favourable and 2 levels that were more favourable. The 5 recommended outcome levels for each goal were assigned numeric values from -2 (the least favourable outcome) to +2 (the most favourable outcome). The expected outcome or goal was assigned 0.

CONTACTS AND LOCATIONS:
Overall Officials: Mintaze Kerem Gunel, PT, PhD, Study Director — Hacettepe University; Zafer Erden, PT, PhD, Study Director — Hacettepe University

IPD SHARING:
Plan to Share IPD: Yes